CLINICAL TRIAL: NCT05750420
Title: Psychological Status and Self-care: a Preliminary Study Involving Patients With Chronic Cardiovascular Disease
Brief Title: Psychological Status and Self-care in Chronic Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: CCM1789
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Anxiety; Depression; Emotional Stress; Quality of Life; Self-care; Chronic Cardiovascular Disease
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There was no intervention, the study was a cross-sectional observational study — Questionnaires for measuring self-care, anxiety, depression, emotinal distress and quality of live were administered to patients with chronic cardiovascular disease

SUMMARY:
This is an observational study aimed at exploring the relationship between psychological status and self-care in patients with chronic cardiovascular disease

DETAILED DESCRIPTION:
400 patients with chronic cardiovascular disease were enrolled in this observational study aiming at exploring the relationship between their psychological status (anxiety, depression, emotional distress and quality of life) and their self-care.

ELIGIBILITY:
Inclusion Criteria:

* Being aged > 18 years old and > 85 years old
* Being diagnosed with a chronic cardiovascular disease
* Being able and willing to sign the Informed Consent Form

Exclusion Criteria:

* Having a cognitive dysfunction or psychotic disorder signaled in the clinical documentation
* Not speaking Italian

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Psychological status and self-care | At the moment of enrollment
  Investigating the relationship between psychological status and self-care in patients with chronic cardiovascular disease

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Monzino Cardiology Center, Milan
  - IRCCS San Gerardo, Monza

IPD SHARING:
Plan to Share IPD: No